CLINICAL TRIAL: NCT00308165
Title: A Phase I Study of Topotecan by Intracerebral Clysis for the Treatment of Recurrent Primary Malignant Brain Tumors
Brief Title: Topotecan by Intracerebral Clysis for Recurrent Primary Malignant Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeffrey N. Bruce (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jeffrey N. Bruce, Edgar M. Housepian Professor of Neurological Surgery Research, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAA4229; R01CA089395 (NIH); NCT00324844 (obsolete NCT alias); NCT00452959 (obsolete NCT alias)
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Results first posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Brain Neoplasms, Primary Malignant
Keywords: Recurrent Primary Malignant Brain Tumors; Brain Tumors; Neoplasms, Brain; Brain Cancer; Brain cancer treatment; Topotecan
MeSH Terms: conditions — Brain Neoplasms | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Topotecan (Experimental): Once a plastic catheter is placed, within 24 hours of placement, the catheter will be connected to a small pump at the bedside, and the convection-enhanced delivery of the Topotecan will begin. The Topotecan will be infused for 4 to 5 days after which time the catheters will simply be pulled out. Patients will be monitored with blood tests and MRI scans during the treatment and at different time periods during the following months.
  Interventions: Procedure: Convection-Enhanced Delivery; Drug: Topotecan

INTERVENTIONS:
Procedure: Convection-Enhanced Delivery — microinfusion pumps to deliver chemotherapy directly into brain tumors
  Other Names: Intracerebral Clysis
Drug: Topotecan — chemotherapeutic drug for the treatment of brain tumors
  Other Names: Hycamtin

SUMMARY:
This study will evaluate the safety and efficacy of a chemotherapeutic drug (topotecan) as it is given directly into brain tumors by a delivery technique called convection-enhanced delivery. This drug has been used for different types of cancer, but in this study it will be given by an experimental delivery technique designed to maximize the amount of drug delivered to the brain tumor and minimize the side effects in other parts of the body.

This study will also evaluate advanced magnetic resonance (MR) imaging techniques.

The study will assess quality of life parameters throughout the follow-up period.

DETAILED DESCRIPTION:
Clinical efficacy with chemotherapy has been discouraging for malignant brain tumors, mostly because of side effects and delivery limitations. Because they are locally invasive and rarely metastasize, malignant gliomas have features that make them uniquely amenable to new strategies of regional drug delivery. Intracerebral clysis (convection-enhanced delivery) is a novel drug delivery strategy that uses a microinfusion pump to establish a pressure gradient in the brain via implanted catheters. The pressure gradient produces convective forces that distribute a therapeutic agent throughout the tumor and surrounding brain tissue.

Non-invasive magnetic resonance imaging (MRI) methods of monitoring drug distribution and treatment response have been developed to maximize the clinical applications and minimize complications associated with treatment risks.

Study participants will be taken to the operating room to have 2 catheters surgically placed into their tumor and surrounding tumor bed. These catheters will then be connected to small infusion pumps which will slowly infuse topotecan continuously over 4-5 days. Patients will have daily MRI scans while in the hospital. Upon completion of the experimental treatment, patients will be discharged and will be followed up in the outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary malignant brain tumor, or a newly diagnosed or recurrent malignant tumor of the brainstem. Patients with tumors of the brain must have been previously treated with external beam radiation. Patients with brainstem gliomas may or may not have been previously treated.
* Patients with a tumor that is stereotactically accessible (MR scan must be obtained within 30 days of enrollment and must demonstrate an enhancing mass without significant mass effect. Tumors must be less than 100 cc in total volume).
* Patients who demonstrate evidence of increasing contrast enhancement on MR or CT imaging while on stable or increasing dose of steroid.
* Patients with a Karnofsky Performance Score of greater than or equal to 60.
* Men and women of child-bearing potential must practice birth control. Women of child bearing potential must have a negative serum or urine pregnancy test within 7 days of study entry.
* Patients must possess the ability to give Informed Consent. Parent or guardian may give informed consent for minors.
* Patients must be willing to and medically capable of undergoing the surgical operation.
* Patients may not be receiving other investigational agents for the treatment of malignant astrocytoma.
* There is no upper age limit. Patients at extreme upper end of the age spectrum will not be automatically excluded, but will be carefully scrutinized to determine their suitability for this procedure.
* Patients must be at least 1 year old to participate in the study.

Exclusion Criteria:

* Patients with diffuse subependymal or cerebrospinal fluid (CSF) disease.
* Patients with tumors involving the cerebellum, or both hemispheres.
* Patients with an active infection requiring treatment or having an unexplained febrile illness.
* Patients who are known HIV positive or who are known positive for Hepatitis B or C virus
* Patients who have received any form of radiation or chemotherapy within 4 weeks of protocol enrollment.
* Patients with systemic diseases which may be associated with unacceptable anesthetic/operative risk.
* Patients who have previously received systemic topotecan for their tumor
* Patients less than 1 year of age
* Patients who are not able to receive an MRI scan

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-03 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bruce, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center Neurological Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Anderson RC, Kennedy B, Yanes CL, Garvin J, Needle M, Canoll P, Feldstein NA, Bruce JN. Convection-enhanced delivery of topotecan into diffuse intrinsic brainstem tumors in children. J Neurosurg Pediatr. 2013 Mar;11(3):289-95. doi: 10.3171/2012.10.PEDS12142. Epub 2012 Dec 14. PMID 23240851

RESULTS

PARTICIPANT FLOW:
Groups:
- Topotecan 0.02 mg/mL: Cohort 1: Patients received 0.02 mg/mL infusion of topotecan through convection-enhanced delivery.
- Topotecan 0.04 mg/mL: Cohort 2: Patients received 0.04 mg/mL infusion of topotecan through convection-enhanced delivery.
- Topotecan 0.0667 mg/mL: Cohort 3: Patients received 0.0667 mg/mL infusion of topotecan through convection-enhanced delivery.
- Topotecan 0.1 mg/mL: Cohort 4: Patients received 0.1 mg/mL infusion of topotecan through convection-enhanced delivery.
- Topotecan 0.133 mg/mL: Cohort 5: Patients received 0.133 mg/mL infusion of topotecan through convection-enhanced delivery.
Period: Dose Level 1: 0.02 mg/mL
Arm/Group | Topotecan 0.02 mg/mL | Topotecan 0.04 mg/mL | Topotecan 0.0667 mg/mL | Topotecan 0.1 mg/mL | Topotecan 0.133 mg/mL
Started | 3 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Level 2: 0.04 mg/mL
Arm/Group | Topotecan 0.02 mg/mL | Topotecan 0.04 mg/mL | Topotecan 0.0667 mg/mL | Topotecan 0.1 mg/mL | Topotecan 0.133 mg/mL
Started | 0 | 3 | 0 | 0 | 0
Completed | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Level 3: 0.0667 mg/mL
Arm/Group | Topotecan 0.02 mg/mL | Topotecan 0.04 mg/mL | Topotecan 0.0667 mg/mL | Topotecan 0.1 mg/mL | Topotecan 0.133 mg/mL
Started | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Level 4: 0.1 mg/mL
Arm/Group | Topotecan 0.02 mg/mL | Topotecan 0.04 mg/mL | Topotecan 0.0667 mg/mL | Topotecan 0.1 mg/mL | Topotecan 0.133 mg/mL
Started | 0 | 0 | 0 | 3 | 0
Completed | 0 | 0 | 0 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Level 5: 0.133 mg/mL
Arm/Group | Topotecan 0.02 mg/mL | Topotecan 0.04 mg/mL | Topotecan 0.0667 mg/mL | Topotecan 0.1 mg/mL | Topotecan 0.133 mg/mL
Started | 0 | 0 | 0 | 0 | 4
Completed | 0 | 0 | 0 | 0 | 4
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topotecan 0.02 mg/mL | Topotecan 0.04 mg/mL | Topotecan 0.0667 mg/mL | Topotecan 0.1 mg/mL | Topotecan 0.133 mg/mL | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 3 | 2 | 3 | 13
  >=65 years | 0 | 1 | 0 | 1 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 0 | 2 | 5
  Male | 2 | 2 | 2 | 3 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Time Frame: During treatment, up to 5 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Topotecan 0.02 mg/mL | Topotecan 0.04 mg/mL | Topotecan 0.0667 mg/mL | Topotecan 0.1 mg/mL | Topotecan 0.133 mg/mL
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 2

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: If 2 participants within a cohort develop dose-limiting toxicity (DLT), the prior dose level is considered the maximum tolerated dose (MTD). Dose-Limiting Toxicities (DLT) will be defined as any new (or increased from baseline) treatment-related (drug and/or device) neurological deficits as exhibited on neurological examination with severity of grade 3 or higher.
Time Frame: During treatment, up to 5 Days
Measure: Number; unit: mg/ml
Arm/Group | Topotecan
Number analyzed (Participants) | 16
mg/ml | 0.1

3. Secondary Outcome: Time to Tumor Progression/Recurrence
Description: Time to tumor progression/recurrence in weeks.
Time Frame: Treatment to progression, Up to 8 years
Population: 1 participant in Cohort 1 died before progression due to disease complications unrelated to treatment. 2 participants in Cohort 5 had not reached progression. These participants were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Topotecan 0.02 mg/mL | Topotecan 0.04 mg/mL | Topotecan 0.0667 mg/mL | Topotecan 0.1 mg/mL | Topotecan 0.133 mg/mL
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 2
Weeks | 70.5 (74.2) | 6.7 (2.3) | 31.7 (6.4) | 36.7 (32.5) | 15.0 (11.3)

4. Secondary Outcome: Time to Death
Description: Time to death measured in weeks
Time Frame: Treatment to Time of Death, Up to 8 Years
Population: Death had not occurred in 1 participant in Cohort 1, 1 participant in Cohort 4, and 2 participants in Cohort 5. These participants were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Topotecan 0.02 mg/mL | Topotecan 0.04 mg/mL | Topotecan 0.0667 mg/mL | Topotecan 0.1 mg/mL | Topotecan 0.133 mg/mL
Number analyzed (Participants) | 2 | 3 | 3 | 2 | 2
weeks | 80 (101.8) | 46 (33.5) | 54 (19.2) | 35.7 (47.8) | 27.3 (28.6)

ADVERSE EVENTS:
Arm/Group | Topotecan 0.02 mg/mL | Topotecan 0.04 mg/mL | Topotecan 0.0667 mg/mL | Topotecan 0.1 mg/mL | Topotecan 0.133 mg/mL
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/3 | 3/3 | 2/3 | 2/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 2/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topotecan 0.02 mg/mL (N=3) | Topotecan 0.04 mg/mL (N=3) | Topotecan 0.0667 mg/mL (N=3) | Topotecan 0.1 mg/mL (N=3) | Topotecan 0.133 mg/mL (N=4)
Parietal syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Upper extremity weakness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes